CLINICAL TRIAL: NCT02253719
Title: Screening for Prevention of Cervical Cancer in HIV-positive and HIV-negative Cambodian Women Using Direct Visualization With Acetic Acid
Brief Title: Cervical Cancer Screening in HIV Positive and Negative Women in Cambodia
Status: Completed | Type: Observational
Sponsor: Sihanouk Hospital Center of HOPE (Other)
Responsible Party: Sponsor
Other Study IDs: SHCH-Cervical Screening-VIA
Record Dates: First submitted 2014-09-17; First posted 2014-10-01 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Cervical Neoplasia; Cervical Cancer
Keywords: cervical neoplasia; cervical cancer'; visual inspection acetic acid; cryotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cryotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HIV positive women: 500 HIV women will be recruited from the hospital's current patient base as well as the community
  Interventions: Procedure: cryotherapy, further biopsy, LEEP, surgery as indicated
- HIV negative women: 500 HIV women will be recruited from the hospital's current patient base as well as the community
  Interventions: Procedure: cryotherapy, further biopsy, LEEP, surgery as indicated

INTERVENTIONS:
Procedure: cryotherapy, further biopsy, LEEP, surgery as indicated — These interventions and their outcomes are not part of this study. However, we will be offering at no charge appropriate treatment for neoplasia or cancer that is diagnosed.

SUMMARY:
The prevalence of cervical neoplasia in Cambodia is not known. There are no screening programs in place. The investigators plan on introducing a screening program based on WHO criteria and utilizing visualization with acetic acid. Patients who are positive will be offered same-day cryotherapy if indicated or will be referred for biopsy, LEEP and hysterectomy as indicated. The planned patient pool for this study is 1000 women, half of whom will be HIV positive (and thus have a presumed higher incidence of cervical neoplasia).

ELIGIBILITY:
Inclusion Criteria:

* female, age 30-49, able to give informed consent

Exclusion Criteria:

* pregnancy, gross cervical mass, prior cervical cancer, unable to give informed consent, prior complete hysterectomy, allergic to acetic acid

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The 1000 women will be recruited from the current patient base of Sihanouk hospital and the surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of cervical neoplasia in HIV positive women | up to 12 months
  500 HIV positive women will be screened for cervical neoplasia using direct visualization with acetic acid
Prevalence of cervical neoplasia in HIV negative women | up to 12 months
  500 HIV negative women will be screened for cervical neoplasia using direct visualization with acetic acid

SECONDARY OUTCOMES:
Treatment of HIV positive women who screen as positive | up to 12 months
  Patients who screen positive will be offered same-day cryotherapy, further diagnostic work-up, and further therapeutic options such as LEEP and hysterectomy as clinically indicated.
Treatment of HIV negative women who screen as positive | up to 12 months
  Patients who screen positive will be offered same-day cryotherapy, further diagnostic work-up, and further therapeutic options such as LEEP and hysterectomy as clinically indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Thay Sovanarra, MD, Principal Investigator — Sihanouk Hospital
Locations (1):
- Sihanouk Hospital, St. 134, Sangkat Vealvong, Khan 7 Makara, Phnom Pehn, Cambodia